CLINICAL TRIAL: NCT06998862
Title: Efficacy of Colchicine in Secondary Prevention of Vascular Events and Renal Progression in Patients With Moderate Chronic Kidney Disease
Brief Title: Colchicine in Chronic Kidney Disease Patients
Acronym: COLCHIREN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FIBHGM-ECNC002-2022; 2023-505868-11-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-04; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Chronic Kidney Disease; Cardiovascular Events
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine treatment (Active Comparator): after randomization, a 0.5 mg tablet of colchicine per day will be administered.
  Interventions: Drug: colchicine treatment in chronic kidney disease patients
- placebo treatment (Placebo Comparator): after randomization 0,25 mg of placebo per day will be administered
  Interventions: Drug: placebo treatment

INTERVENTIONS:
Drug: colchicine treatment in chronic kidney disease patients — colchicine treatment 0.5 mg/day
  Arms: Colchicine treatment
Drug: placebo treatment — placebo treatment 1 pill/day
  Arms: placebo treatment

SUMMARY:
The ColchiRen study is a phase 3, controlled, prospective, randomized, double-blind, and multicenter clinical trial. Its main objective is to demonstrate the benefit of low-dose colchicine treatment in secondary prevention of cardiovascular events in patients with moderate CKD. As a secondary objective, it aims to explore the potential beneficial anti-inflammatory effect on the progression of CKD.

DETAILED DESCRIPTION:
A total of 744 patients will be included (50% in each branch), and the follow-up time of the study will be three years.

EXPLORATORY PARAMETERS

* Analytical parameters in blood:

  * Hemogram: hemoglobin, erythrocyte sedimentation rate.
  * Biochemistry: creatinine, glomerular filtration rate estimated by CKD-EPI, glucose, triglycerides, total cholesterol, HDL-cholesterol, LDL-cholesterol, uric acid, C-reactive protein, fibrinogen, glycosylated hemoglobin.
* Analytical parameter in urine: albumin/creatinine ratio in first morning urine.
* Parameters in samples centralized in the Renal Pathophysiology Laboratory: array including more than 40 molecules that promote and inhibit inflammation and fibrosis; measurement of ACE and ACE2.
* Cardiovascular events defined as one of the following:

  * Cardiovascular death.
  * Acute coronary syndrome.
  * Angina requiring hospitalization.
  * Coronary revascularization.
  * Transient ischemic attack or noncardioembolic ischemic stroke.
  * Peripheral vascular disease, defined as acute peripheral arterial embolism or ischemia, or need for amputation or percutaneous surgical revascularization.
* Renal event, defined as one of the following:

  * 40% decrease in glomerular filtration rate estimated by CKD-EPI with respect to baseline.
  * Doubling of serum creatinine above baseline.
  * Persistent drop in glomerular filtration rate estimated by CKD-EPI below 15 mL/min/1.73m2.
  * Need for renal replacement therapy

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 99 years. Moderate chronic kidney disease, defined as an estimated glomerular filtration rate (eGFR) by the CKD-EPI formula between 30 and 59 mL/min/1.73 m².

History of a previous cardiovascular event:

Acute coronary syndrome. Admission for angina pectoris. Transient ischemic attack or non-cardioembolic ischemic stroke. Coronary revascularization. Peripheral vasculopathy, defined as: embolism or acute peripheral arterial ischemia, or the need for amputation or surgical revascularization.

Finding of coronary artery disease on imaging test.

Exclusion Criteria:

* History of allergy or intolerance to colchicine or any of its excipients (dihydrate calcium hydrogen phosphate, microcrystalline cellulose, anhydrous colloidal silica, magnesium stearate).
* Current treatment with colchicine, or within the month prior to inclusion.
* Hospital admission for any cause within the 3 months prior to study inclusion.
* Active malignant neoplasm (except non-melanoma skin cancer or carcinoma in situ). Patients with a history of malignant neoplasm who have remained disease-free for the past 3 years may be included.
* Uncontrolled or symptomatic chronic inflammatory disease (rheumatoid arthritis, systemic lupus erythematosus, Crohn's disease, ulcerative colitis, etc.).
* Active infection with hepatitis B virus, hepatitis C virus, or human immunodeficiency virus.
* Liver cirrhosis of any cause, grade B or C according to Child-Pugh.
* Immunosuppressive treatment within the 12 weeks prior to study inclusion.
* Chronic treatment with non-steroidal anti-inflammatory drugs (NSAIDs).
* Poorly controlled hypertension (>160/90 mmHg) at the time of inclusion.
* Pregnancy and breastfeeding at the time of inclusion. Contraceptive methods are required for women of reproductive age. Women with no capacity for pregnancy are considered to be those with:

History of hysterectomy, bilateral salpingectomy, bilateral oophorectomy, or bilateral tubal ligation.

Documented infertility. Postmenopausal women, defined as amenorrhea for more than 12 months without other medical cause. In case of doubt, confirmation with elevated follicle-stimulating hormone (FSH) levels is recommended.

Women of reproductive capacity must use a method of contraception with proven effectiveness until 8 weeks after the end of the study. Acceptable methods include:

Intrauterine device (IUD) placement at least 6 weeks before study inclusion. Hormonal contraception with progestogens only, associated with ovulation inhibition: oral, injectable, or implantable, at least 6 weeks before study inclusion.

Progestin-releasing intrauterine system (IUS) at least 6 weeks before study inclusion.

Combined hormonal contraception (containing estrogen and progestogens) associated with ovulation inhibition: oral, intravaginal, transdermal, at least 6 weeks before study inclusion.

Other contraceptive methods (sexual abstinence, barrier methods, spermicides, etc.) are not considered acceptable for participation in this study

* Gastric ulcer
* thrombocytopenia <50,000 cells/μL during the month prior to inclusion
* Neutropenia defined as <1500 cells/mcL during the month prior to inclusion.
* Anemia defined as hemoglobin <10.5 g/dL during the month prior to inclusion.
* History of aplastic anemia diagnosed through bone marrow biopsy.
* Treatment with CYP3A4 inhibitors and/or P-glycoprotein inhibitors (antivirals, azole antifungals, aminoglycosides, cyclosporine) in the month prior to their inclusion in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — all
Enrollment: 744 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular events | from enrollment to the end of treamtent at three years
  Incidence of the primary event consisting of death due to cardiovascular causes; acute coronary syndrome; angina requiring hospitalization; coronary revascularization; transient ischemic attack or non-cardioembolic ischemic stroke; or peripheral vasculopathy, defined as embolism or acute peripheral arterial ischemia, or the need for amputation or surgical or percutaneous revascularization."

SECONDARY OUTCOMES:
cardiovascular death | from enrollment to the end of treamtent at three years
  Incidence of death due to cardiovascular causes.
Acute coronary syndrome | from enrollment to the end of treamtent at three years
  Incidence of acute coronary syndrome
Angina pectoris | from enrollment to the end of treamtent at three years
  Incidence of hospitalization for angina pectoris.
stroke | from enrollment to the end of treamtent at three years
  Incidence of transient ischemic attack or non-cardioembolic ischemic stroke.
Peripheral vasculopathy | from enrollment to the end of treamtent at three years
  Incidence of peripheral vasculopathy, defined as embolism or acute peripheral arterial ischemia, or the need for amputation or surgical revascularization.
renal disease progression | from enrollment to the end of treamtent at three years
  Individual and combined incidence of renal events:
  A 40% decrease in estimated glomerular filtration rate (eGFR) by CKD-EPI compared to baseline, doubling of serum creatinine over its baseline level, Persistent decline in estimated glomerular filtration rate (eGFR) by CKD-EPI below 15 mL/min/1.73 m² or need for sustained renal replacement therapy.
effect of colchcine treatment on inflammation and fibrosis parameters | from enrollment to the end of treatment at three years
  At the baseline, annual and final visits of the study, an additional blood sample will be obtained, which will be frozen at -80º and sent for centralized analysis at the Renal Physiopathology Laboratory of the Hospital General Universitario Gregorio Marañón. The measurement will be performed using cytokine arrays (Human Inflammation Array, RayBiotech®) with which the measurement of 40 inflammatory/profibrotic and anti-inflammatory factors is contemplated, including among others: TNFα, TNFβ, IL2, IL6, IL7, IL1α, IL1β, IL17A RANTES, ICAM-1, TIMP-1, TIMP-2, GCSF and M-CSF.
Security | from enrollment to the end of treatment at three years
  Incidence of adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario Gregorio Marañon, Madrid, Madrid, Spain